CLINICAL TRIAL: NCT03601832
Title: Phase I/II Study of 4-D Navigated Non-invasive Radiosurgical Ablation of Ventricular Tachycardia
Brief Title: Non-invasive Ablation of Ventricular Tachycardia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Ostrava (Other)
Collaborators: University of Ostrava (Other); Hospital Podlesi (Other); Hospital Nový Jičín (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NIRA-VT; 18/RVO-FNOs/2018 (Other Grant/Funding Number: University Hospital Ostrava)
Record Dates: First submitted 2018-05-18; First posted 2018-07-26 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Ventricular Tachycardia
Keywords: scar-related; ventricular tachycardia; substrate ablation; stereotactic radiosurgery; functional radiosurgery; 4D navigation
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Intervention Model Description: All patients enroled in the study are allocated to one group with 4-D navigated stereotactic radiosurgical ablation.
Masking Description: No masking in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 4-D navigated stereotactic radiosurgical ablation (Experimental): The patients enroled to this arm of the study will undergo 4-D navigated stereotactic radiosurgical ablation.
  Interventions: Procedure: 4-D navigated stereotactic radiosurgical ablation

INTERVENTIONS:
Procedure: 4-D navigated stereotactic radiosurgical ablation — 4-D Navigated Non-invasive radiosurgical ablation of ventricular tachycardia in patients with sustained monomorphic ventricular tachycardia/tachycardias after myocardial infarction.

SUMMARY:
Phase I/II study of 4-D Navigated Non-invasive radiosurgical ablation of ventricular tachycardia (NIRA-VT).

DETAILED DESCRIPTION:
The goal of this project dealing with 4D-navigated substrate ablation is to evaluate the feasibility and safety of elimination of the scar-related monomorphic ventricular tachycardia (VT) or tachycardias by stereotactic radiosurgical ablation that is completely non-invasive. The arrhythmic substrate is defined as the scar after myocardial infarction (MI) described by transthoracic echocardiography (TTE) and specified by PET-CT or MRI. All sustained monomorphic VT induced by programmed ventricular stimulation via implanted ICD (Implantable Cardioverter Defibrillator) will be analyzed using body surface ECG mapping. The target volume for stereotactic radiosurgical ablation (single dose of 25 Gy) will be based on accordance between a post-infarction scar (PET-CT or MRI imaging) and arrhythmic substrate (body surface ECG mapping).

ELIGIBILITY:
Inclusion Criteria:

* history of sustained monomorphic VT or termination of monomorphic VT by ICD (appropriate therapy) during previous 6 months prior to enrollment
* implantation ICD
* inducibility at least one of monomorphic ventricular tachycardia by ICD during EP study with programmed ventricular stimulation
* history of myocardial infarction (MI)
* left ventricular scar and decreased systolic function of the left ventricle (ejection fraction of left ventricle less than 40%) based on transthoracic ultrasound
* stable chronic heart failure (NYHA II-III)
* older than 18 years
* signed an IRB approved written informed consent document.
* failed at least one invasive catheter ablation procedure or have a contraindication to a catheter ablation procedure

Exclusion Criteria:

* acute myocardial infarction
* chronic heart failure NYHA IV
* channelopathy
* reversible cause of VT (e.g. ionic dysbalance, intoxications)
* pregnancy or breastfeeding
* history of chest radiotherapy
* arrhythmic substrate larger than 100 ccm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Composite of death | 90 days
  Composite of death occurring at any time after treatment or arrhythmic storm (three or more documented episodes of VT within 24 hours) or appropriate ICD therapy (both shock and pacing) after a 90-day treatment period. 90-day treatment period was imposed to exclude nonfatal outcomes that might occur during acute radiation reaction. Moreover, functional radiosurgery has 90% success rate after 3 months.
Acute radiation-induced events | 18 months
  Acute radiation-induced events (within 3 months after treatment) according to CTCAE 4.0. Major concern will be on radiation myocarditis, pericarditis and pneumonitis/fibrosis. Needs of antiemetic drugs will be recorded.
Late radiation-induced effects | 18 months
  Late radiation-induced effects (after 3 months after treatment) according to CTCAE 4.0. Major concern will be on radiation myocarditis, pericarditis and pneumonitis/fibrosis. Needs of antiemetic drugs will be recorded.

SECONDARY OUTCOMES:
Time to death at any time | 18 months
Time to arrhythmic storm | 90 days
  Time to arrhythmic storm (three or more documented episodes of VT within 24 hours) at any time and after 90-day treatment period.
Time to appropriate ICD shock | 90 days
  Time to appropriate ICD shock at any time and after 90-day treatment period.
Time to appropriate antitachycardial pacing by ICD | 90 days
  Time to appropriate antitachycardial pacing by ICD at any time and after 90-day treatment period.
Hospitalization due to VT | 18 months
Hospitalization due to chronic heart failure | 18 months
Quality of life measured with EQ-5D questionnaire | 18 months
  Quality of life measurement using a standardised tool named EQ-5D. EQ-5D is a standardised instrument in the form of a questionnaire developed by the EuroQol Group as a measure of health-related quality of life that can be used in a wide range of health conditions and treatments. The EQ-5D instrument consists of a descriptive system and the EuroQol-visual analogue scales (EQ VAS). The quality of life is measured in 5 dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, extreme problems. The higher the score achieved, the higher the quality of life of the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Jakub Cvek, Ing.,MD,Ph.D., Principal Investigator — University Hospital Ostrava
Locations (3):
- Czechia (3):
  - Hospital Nový Jičín, Nuclear Medicine - PET/CT, Nový Jičín, Moravian-Silesian Region
  - University Hospital Ostrava, Ostrava, Moravian-Silesian Region
  - Hospital Podlesí, Třinec, Moravian-Silesian Region

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Connolly SJ, Hallstrom AP, Cappato R, Schron EB, Kuck KH, Zipes DP, Greene HL, Boczor S, Domanski M, Follmann D, Gent M, Roberts RS. Meta-analysis of the implantable cardioverter defibrillator secondary prevention trials. AVID, CASH and CIDS studies. Antiarrhythmics vs Implantable Defibrillator study. Cardiac Arrest Study Hamburg . Canadian Implantable Defibrillator Study. Eur Heart J. 2000 Dec;21(24):2071-8. doi: 10.1053/euhj.2000.2476. PMID 11102258
- [Background] Moss AJ, Zareba W, Hall WJ, Klein H, Wilber DJ, Cannom DS, Daubert JP, Higgins SL, Brown MW, Andrews ML; Multicenter Automatic Defibrillator Implantation Trial II Investigators. Prophylactic implantation of a defibrillator in patients with myocardial infarction and reduced ejection fraction. N Engl J Med. 2002 Mar 21;346(12):877-83. doi: 10.1056/NEJMoa013474. Epub 2002 Mar 19. PMID 11907286
- [Background] Poole JE, Johnson GW, Hellkamp AS, Anderson J, Callans DJ, Raitt MH, Reddy RK, Marchlinski FE, Yee R, Guarnieri T, Talajic M, Wilber DJ, Fishbein DP, Packer DL, Mark DB, Lee KL, Bardy GH. Prognostic importance of defibrillator shocks in patients with heart failure. N Engl J Med. 2008 Sep 4;359(10):1009-17. doi: 10.1056/NEJMoa071098. PMID 18768944
- [Background] Sapp JL, Wells GA, Parkash R, Stevenson WG, Blier L, Sarrazin JF, Thibault B, Rivard L, Gula L, Leong-Sit P, Essebag V, Nery PB, Tung SK, Raymond JM, Sterns LD, Veenhuyzen GD, Healey JS, Redfearn D, Roux JF, Tang AS. Ventricular Tachycardia Ablation versus Escalation of Antiarrhythmic Drugs. N Engl J Med. 2016 Jul 14;375(2):111-21. doi: 10.1056/NEJMoa1513614. Epub 2016 May 5. PMID 27149033
- [Background] Mallidi J, Nadkarni GN, Berger RD, Calkins H, Nazarian S. Meta-analysis of catheter ablation as an adjunct to medical therapy for treatment of ventricular tachycardia in patients with structural heart disease. Heart Rhythm. 2011 Apr;8(4):503-10. doi: 10.1016/j.hrthm.2010.12.015. Epub 2010 Dec 13. PMID 21147263
- [Background] Tung R, Michowitz Y, Yu R, Mathuria N, Vaseghi M, Buch E, Bradfield J, Fujimura O, Gima J, Discepolo W, Mandapati R, Shivkumar K. Epicardial ablation of ventricular tachycardia: an institutional experience of safety and efficacy. Heart Rhythm. 2013 Apr;10(4):490-8. doi: 10.1016/j.hrthm.2012.12.013. Epub 2012 Dec 11. PMID 23246598
- [Background] Di Biase L, Santangeli P, Burkhardt DJ, Bai R, Mohanty P, Carbucicchio C, Dello Russo A, Casella M, Mohanty S, Pump A, Hongo R, Beheiry S, Pelargonio G, Santarelli P, Zucchetti M, Horton R, Sanchez JE, Elayi CS, Lakkireddy D, Tondo C, Natale A. Endo-epicardial homogenization of the scar versus limited substrate ablation for the treatment of electrical storms in patients with ischemic cardiomyopathy. J Am Coll Cardiol. 2012 Jul 10;60(2):132-41. doi: 10.1016/j.jacc.2012.03.044. PMID 22766340
- [Background] Jais P, Maury P, Khairy P, Sacher F, Nault I, Komatsu Y, Hocini M, Forclaz A, Jadidi AS, Weerasooryia R, Shah A, Derval N, Cochet H, Knecht S, Miyazaki S, Linton N, Rivard L, Wright M, Wilton SB, Scherr D, Pascale P, Roten L, Pederson M, Bordachar P, Laurent F, Kim SJ, Ritter P, Clementy J, Haissaguerre M. Elimination of local abnormal ventricular activities: a new end point for substrate modification in patients with scar-related ventricular tachycardia. Circulation. 2012 May 8;125(18):2184-96. doi: 10.1161/CIRCULATIONAHA.111.043216. Epub 2012 Apr 4. PMID 22492578
- [Background] Tzou WS, Frankel DS, Hegeman T, Supple GE, Garcia FC, Santangeli P, Katz DF, Sauer WH, Marchlinski FE. Core isolation of critical arrhythmia elements for treatment of multiple scar-based ventricular tachycardias. Circ Arrhythm Electrophysiol. 2015 Apr;8(2):353-61. doi: 10.1161/CIRCEP.114.002310. Epub 2015 Feb 13. PMID 25681389
- [Background] Chang SD, Main W, Martin DP, Gibbs IC, Heilbrun MP. An analysis of the accuracy of the CyberKnife: a robotic frameless stereotactic radiosurgical system. Neurosurgery. 2003 Jan;52(1):140-6; discussion 146-7. doi: 10.1097/00006123-200301000-00018. PMID 12493111
- [Background] Fariselli L, Marras C, De Santis M, Marchetti M, Milanesi I, Broggi G. CyberKnife radiosurgery as a first treatment for idiopathic trigeminal neuralgia. Neurosurgery. 2009 Feb;64(2 Suppl):A96-101. doi: 10.1227/01.NEU.0000341714.55023.8F. PMID 19165081
- [Background] Regis J, Tuleasca C, Resseguier N, Carron R, Donnet A, Gaudart J, Levivier M. Long-term safety and efficacy of Gamma Knife surgery in classical trigeminal neuralgia: a 497-patient historical cohort study. J Neurosurg. 2016 Apr;124(4):1079-87. doi: 10.3171/2015.2.JNS142144. Epub 2015 Sep 4. PMID 26339857
- [Background] Gianni C, Mohanty S, Trivedi C, Di Biase L, Al-Ahmad A, Natale A, David Burkhardt J. Alternative Approaches for Ablation of Resistant Ventricular Tachycardia. Card Electrophysiol Clin. 2017 Mar;9(1):93-98. doi: 10.1016/j.ccep.2016.10.006. Epub 2016 Dec 24. PMID 28167089
- [Background] Cuculich PS, Schill MR, Kashani R, Mutic S, Lang A, Cooper D, Faddis M, Gleva M, Noheria A, Smith TW, Hallahan D, Rudy Y, Robinson CG. Noninvasive Cardiac Radiation for Ablation of Ventricular Tachycardia. N Engl J Med. 2017 Dec 14;377(24):2325-2336. doi: 10.1056/NEJMoa1613773. PMID 29236642